CLINICAL TRIAL: NCT01130844
Title: A Phase 1, Multicenter, Open-label Study to Determine the Safety and Pharmacokinetics of MMX Mesalamine Following Administration in Children and Adolescents With Ulcerative Colitis
Brief Title: Safety and Pharmacokinetics of MMX Mesalamine in Children and Adolescents With Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SPD476-112; 2011-000164-10 (EudraCT Number)
Record Dates: First submitted 2010-05-20; First posted 2010-05-26 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MMX Mesalamine (30mg/kg) (Experimental)
  Interventions: Drug: MMX Mesalamine
- MMX Mesalamine (60 mg/kg) (Experimental)
  Interventions: Drug: MMX Mesalamine
- MMX Mesalamine (100 mg/kg) (Experimental)
  Interventions: Drug: MMX Mesalamine

INTERVENTIONS:
Drug: MMX Mesalamine — 30 mg/kg/day of MMX Mesalamine tablets, dosed once daily for 7 days.
  Other Names: Lialda, SPD476
  Arms: MMX Mesalamine (30mg/kg)
Drug: MMX Mesalamine — 60 mg/kg/day of MMX Mesalamine tablets, dosed once daily for 7 days.
  Other Names: Lialda, SPD476
  Arms: MMX Mesalamine (60 mg/kg)
Drug: MMX Mesalamine — 100 mg/kg/day of MMX Mesalamine tablets, dosed once daily for 7 days.
  Other Names: Lialda, SPD476
  Arms: MMX Mesalamine (100 mg/kg)

SUMMARY:
The purpose of this study is to determine the safety and pharmacokinetics of MMX mesalamine following administration in children and adolescents with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 5-17 years, with appropriately obtained informed consent and assent.
2. Subject has a documented history of ulcerative colitis for at least 3 months.
3. Subjects who are currently on 5-ASA or product(s) containing or metabolized to mesalamine must have been on a stable regimen for at least 4 weeks prior to first dose of investigational medicinal product.
4. Subjects who are not currently on a drug regimen, or on a 5-ASA or product containing or metabolized to mesalamine, must have been on a stable regimen for at least 4 weeks prior to first dose at least 4 weeks prior first dose of investigational medicinal product.
5. Body weight of 18kg-82kg inclusive.

Exclusion Criteria:

1. Current or recurrent disease (eg cardiovascular, renal, liver, malignancy or other conditions) that could affect the colon, the action, absorption or disposition of the IMP, or clinical or laboratory assessments with the exception of their existing ulcerative colitis.
2. Ulcerative Colitis known to be confined to the rectum (isolated rectal proctitis).
3. Any history of hepatic impairment or moderate to severe renal impairment.
4. The use of systemic or rectal steroids within the last 4 weeks, immunomodulators within the last 6 weeks, biologics within 6 months, antibiotic use within the last 7 days prior to the first dose of investigational medicinal product.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2010-10-08 (Actual); Primary Completion 2013-06-27 (Actual); Study Completion 2013-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (19):
- United States (6):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - University of California, San Francisco, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - University of Maryland Medical Center for Children, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
- Royal Children's Hospital Melbourne, Parkville, Victoria, Australia
- Poland (5):
  - Klinika Pediatrii Gastroenterologii i Zywienia, Uniwersytecki Szpital Dzieciecy w Krakowie, Wieliczka, Krakow
  - Klinika Gastroenterolofii Pediatrii, Instytut Centrum Zdrowia Matki Polki, Lodz
  - Klinika Pediatrii Dzieciecy Szpital Kliniczny im prof Antoniego Gebali, Lublin
  - Kliniczny Oddzial Pediatrii z Pododdzialem Neurologii Dzieciecej Szpital Wojewodzki, Rzeszów
  - Oddzial Gastroenterologii i Hepatologii, Instytut Pomnik-Centrum Zdrowia Dziecka, Warsaw
- Slovakia (3):
  - Univerzitna nemocnica Martin, Martin, Kollarova 2
  - DFNsP Banska Bystrica, Banská Bystrica
  - Gastroenterologicka ambulancia, Bratislava
- United Kingdom (4):
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust/Royal London Hospital, London
  - Somers Clinical Research Facility/Great Ormond Street Hospital, London
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Cuffari C, Pierce D, Korczowski B, Fyderek K, Van Heusen H, Hossack S, Wan H, Edwards AY, Martin P. Randomized clinical trial: pharmacokinetics and safety of multimatrix mesalamine for treatment of pediatric ulcerative colitis. Drug Des Devel Ther. 2016 Feb 4;10:593-607. doi: 10.2147/DDDT.S95316. eCollection 2016. PMID 26893546

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MMX Mesalamine (30mg/kg) | MMX Mesalamine (60 mg/kg) | MMX Mesalamine (100 mg/kg)
Started | 21 | 22 | 9
Completed | 21 | 22 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MMX Mesalamine (30mg/kg) | MMX Mesalamine (60 mg/kg) | MMX Mesalamine (100 mg/kg) | Total
Number analyzed (Participants) | 21 | 22 | 9 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.0 (2.88) | 13.9 (2.59) | 10.6 (3.28) | 13.3 (3.06)
Age, Customized [Count of Participants; unit: Participants]
  5 to 17 years, inclusive | 21 | 22 | 9 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 5 | 30
  Male | 7 | 11 | 4 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 4 | 1 | 8
  Slovakia | 2 | 1 | 0 | 3
  Poland | 16 | 17 | 8 | 41

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of MMX Mesalamine (5-ASA) at Steady State
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: 2, 4, 6, 9, 12, 16, and 24 hours post-dose on day 7
Population: The Pharmacokinetic Set (PKS) consisted of all subjects in the Safety Analysis Set who generated sufficient plasma samples to allow reliable determination of Cmax and AUC. The Safety Analysis Set consisted of subjects who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Measure: Mean (Standard Deviation); unit: ug*h/L
Arm/Group | MMX Mesalamine (30mg/kg) | MMX Mesalamine (60 mg/kg) | MMX Mesalamine (100 mg/kg)
Number analyzed (Participants) | 21 | 22 | 9
ug*h/L | 21411 (11081) | 46173 (22864) | 49213 (17664)

2. Secondary Outcome: Percentage of Dose Absorbed For MMX Mesalamine (5-ASA) in Urine at Steady State
Description: The percentage of the dose absorbed was calculated as: 100 x (Xu0-24h 5-ASA + [0.7847* Xu0-24h Ac-5-ASA])/dose, where 0.7847 is the ratio of the molecular weight of 5-ASA (153.14) to the molecular weight of Ac-5-ASA (195.15). Xu0-24h is equal to the cumulative amount recovered in urine in the time interval of 0 to 24 hours.
Time Frame: Over a 24-hour period starting on day 7
Population: PKS
Measure: Mean (Standard Deviation); unit: percentage of dose absorbed
Arm/Group | MMX Mesalamine (30mg/kg) | MMX Mesalamine (60 mg/kg) | MMX Mesalamine (100 mg/kg)
Number analyzed (Participants) | 21 | 22 | 9
percentage of dose absorbed | 29.4 (14.5) | 27.0 (13.5) | 22.1 (13.6)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of MMX Mesalamine (5-ASA) at Steady State
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: Over a 24-hour period starting on day 7
Population: PKS
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | MMX Mesalamine (30mg/kg) | MMX Mesalamine (60 mg/kg) | MMX Mesalamine (100 mg/kg)
Number analyzed (Participants) | 21 | 22 | 9
ug/L | 1884 (1018) | 3825 (1979) | 4314 (2602)

4. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of MMX Mesalamine (5-ASA) at Steady State
Description: Tmax is the time after administration of a drug when the maximum plasma concentration in the body is reached.
Time Frame: Over a 24-hour period starting on day 7
Population: PKS
Measure: Median (Full Range); unit: hours
Arm/Group | MMX Mesalamine (30mg/kg) | MMX Mesalamine (60 mg/kg) | MMX Mesalamine (100 mg/kg)
Number analyzed (Participants) | 21 | 22 | 9
hours | 6.00 [0.00 to 24.0] | 8.98 [0.00 to 24.0] | 1.98 [0.00 to 24.0]

5. Primary Outcome: Total Body Clearance (CL) of MMX Mesalamine (5-ASA) at Steady State
Description: Clearance of a substance from the blood by the kidneys.
Time Frame: Over a 24-hour period starting on day 7
Population: PKS
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | MMX Mesalamine (30mg/kg) | MMX Mesalamine (60 mg/kg) | MMX Mesalamine (100 mg/kg)
Number analyzed (Participants) | 21 | 22 | 9
L/h | 6.48 (2.99) | 5.94 (2.95) | 4.95 (2.07)

6. Primary Outcome: AUC of MMX Mesalamine Major Metabolite (Ac-5-ASA) at Steady State
Time Frame: 2, 4, 6, 9, 12, 16, and 24 hours post-dose on day 7
Population: PKS
Measure: Mean (Standard Deviation); unit: ug*h/L
Groups:
- MMX Mesalamine Metabolite (30mg/kg): MMX Mesalamine: 30 mg/kg/day of MMX Mesalamine tablets, dosed once daily for 7 days.
- MMX Mesalamine Metabolite (60 mg/kg): MMX Mesalamine: 60 mg/kg/day of MMX Mesalamine tablets, dosed once daily for 7 days.
- MMX Mesalamine Metabolite (100 mg/kg): MMX Mesalamine: 100 mg/kg/day of MMX Mesalamine tablets, dosed once daily for 7 days.
Arm/Group | MMX Mesalamine Metabolite (30mg/kg) | MMX Mesalamine Metabolite (60 mg/kg) | MMX Mesalamine Metabolite (100 mg/kg)
Number analyzed (Participants) | 21 | 22 | 9
ug*h/L | 30942 (13743) | 58119 (22729) | 63067 (21752)

7. Primary Outcome: Cmax of MMX Mesalamine Major Metabolite (Ac-5-ASA) at Steady State
Time Frame: Over a 24-hour period starting on day 7
Population: PKS
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | MMX Mesalamine Metabolite (30mg/kg) | MMX Mesalamine Metabolite (60 mg/kg) | MMX Mesalamine Metabolite (100 mg/kg)
Number analyzed (Participants) | 21 | 22 | 9
ug/L | 2396 (1217) | 4113 (1641) | 4968 (2911)

8. Primary Outcome: Tmax of MMX Mesalamine Major Metabolite (Ac-5-ASA) at Steady State
Time Frame: Over a 24-hour period starting on day 7
Population: PKS
Measure: Median (Full Range); unit: hours
Arm/Group | MMX Mesalamine Metabolite (30mg/kg) | MMX Mesalamine Metabolite (60 mg/kg) | MMX Mesalamine Metabolite (100 mg/kg)
Number analyzed (Participants) | 21 | 22 | 9
hours | 9.00 [0.00 to 24.0] | 7.48 [0.00 to 24.0] | 1.98 [0.00 to 24.0]

9. Primary Outcome: CL of MMX Mesalamine Major Metabolite (Ac-5-ASA) at Steady State
Time Frame: Over a 24-hour period starting on day 7
Population: PKS
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | MMX Mesalamine Metabolite (30mg/kg) | MMX Mesalamine Metabolite (60 mg/kg) | MMX Mesalamine Metabolite (100 mg/kg)
Number analyzed (Participants) | 21 | 22 | 9
L/h | 16.2 (6.72) | 12.2 (4.43) | 10.0 (4.36)

10. Secondary Outcome: Cumulative Amount of MMX Mesalamine (5-ASA) Recovered in Urine at Steady State
Time Frame: Over a 24-hour period starting on day 7
Population: PKS
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | MMX Mesalamine (30mg/kg) | MMX Mesalamine (60 mg/kg) | MMX Mesalamine (100 mg/kg)
Number analyzed (Participants) | 21 | 22 | 9
mg | 162 (132) | 298 (221) | 235 (121)

11. Secondary Outcome: Cumulative Amount of MMX Mesalamine Major Metabolite (Ac-5-ASA) Recovered in Urine at Steady State
Time Frame: Over a 24-hour period starting on day 7
Population: PKS
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | MMX Mesalamine Metabolite (30mg/kg) | MMX Mesalamine Metabolite (60 mg/kg) | MMX Mesalamine Metabolite (100 mg/kg)
Number analyzed (Participants) | 21 | 22 | 9
mg | 532 (411) | 708 (341) | 593 (251)

ADVERSE EVENTS:
Arm/Group | MMX Mesalamine (30mg/kg) | MMX Mesalamine (60 mg/kg) | MMX Mesalamine (100 mg/kg)
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/9
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.